CLINICAL TRIAL: NCT06881004
Title: Establishment and Evaluation of Clinical Classification and Surgical Decision-making System for Biliary Dilatation：a National Special Disease Cohort Study in China
Brief Title: Biliary Dilatation National Special Disease Cohort in China
Status: Recruiting | Type: Observational
Sponsor: Beijing Tsinghua Chang Gung Hospital (Other)
Responsible Party: Principal Investigator, Shuo Jin, Associate Chief Physician, Beijing Tsinghua Chang Gung Hospital
Other Study IDs: 24640-0-01
Record Dates: First submitted 2025-03-11; First posted 2025-03-18 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Choledochal Cyst
Keywords: Biliary dilatation; Cohort study; Clinical database; Surgical treatment; Long-term outcome
MeSH Terms: conditions — Choledochal Cyst

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Retrospective cohort: This cohort retrospectively collects all available clinical data and prognostic information of all patients who were previously diagnosed with biliary dilatation in the participating centers, and compares the various outcome indicators of two groups or multiple groups.
- Prospective cohort: This cohort prospectively enrolls all patients with a clear diagnosis of biliary dilatation in each participating center, tracks and observes them for a certain period of time, and compares the various outcome indicators of two groups or multiple groups. Additionally, it conducts prospective follow-ups on the patients in the retrospective cohort.

SUMMARY:
This study is a multicenter, bidirectional cohort study aimed at continuously enrolling patients with biliary dilatation from 25 medical centers in China. It will collect comprehensive life-cycle data from the cohort to establish a Chinese cohort for bile duct dilatation. Based on this cohort, the study seeks to clarify the epidemiological characteristics, pathological features, standard classification, disease progression, cancer risk, and optimal timing for surgical intervention in patients with bile duct dilatation. Additionally, it will compare the perioperative risks, long-term outcomes, and quality of life among different types of patients (including Todani types I, IVa, and V) following surgical treatment, to establish standardized surgical treatment strategies for each type.

DETAILED DESCRIPTION:
Biliary Dilatation(BD) is a complex benign biliary disorder prevalent in East Asia, for which surgical resection remains the sole curative approach necessitating prompt intervention upon diagnosis. Nevertheless, critical aspects including disease subtyping, standardized surgical management protocols, and prognostic determinants remain inadequately defined. This multicenter ambidirectional cohort study aims to consecutively enroll BD patients across 25 tertiary medical centers in China, systematically collecting comprehensive life-cycle data encompassing demographic profiles, clinical baseline characteristics, laboratory/imaging findings, biliary-specific biomarkers, and longitudinal follow-up records to establish a nationally representative Chinese BD cohort. Building upon this cohort, the study objectives are structured as follows:

1. Establishment and Maintenance: To construct and perpetually update a multicenter clinical database for BD research in China, ensuring data integrity and accessibility.
2. Age-Stratified Comparative Analysis: To delineate and contrast the differential patterns of disease progression, surgical decision-making paradigms, and postoperative surveillance strategies between adult and pediatric BD populations.
3. Natural History Characterization: To elucidate disease trajectories, morphological evolution, comorbidity progression, malignant transformation risks, and evidence-based surgical indications/timing in non-operated asymptomatic BD patients.
4. Therapeutic Standardization: To define optimal surgical modalities (with emphasis on Todani classification types I, IVa, and V) and critically evaluate the efficacy-safety profile of standardized operative approaches through multidimensional outcome assessments.
5. Quality-of-Life Quantification: To systematically evaluate postoperative quality of life (QoL) metrics across BD subtypes and identify modifiable determinants influencing long-term patient-reported outcomes.
6. Epidemiological Benchmarking: To synthesize epidemiological patterns, establish evidence-based clinical endpoints for surgical interventions, and define reference standards for treatment-related risks and QoL benchmarks in standardized BD management.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have been definitive diagnosed with biliary dilation.
2. Patients aged between 0 and 80 years old, regardless of gender.
3. In line with the principle of informed consent: For the retrospective cohort of biliary dilation, exemption from signing the informed consent form is applied for, while for the prospective cohort, signing the informed consent form is required.

Exclusion Criteria:

* None

Max Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with a definitive diagnosis of biliary dilation in the participating centers will be included.
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2025-03-19 (Actual); Primary Completion 2035-03-31 (Estimated); Study Completion 2035-03-31 (Estimated)

PRIMARY OUTCOMES:
Long-term complications rate | After 30 or 90 days of surgery
  For patients who have undergone surgical treatment, the occurrences of long-term postoperative complications include recurrent cholangitis, pancreatitis, bile duct stones, liver failure, and other such conditions.

SECONDARY OUTCOMES:
Malignant transformation rate | through study completion, an average of 10 year
  The occurrence of malignant transformation associated with bile duct dilatation
Perioperative complication rate | Within 30 or 90 days postoperatively
  The occurrence of perioperative complications, including bile leakage, pancreatic leakage, liver failure, bacteremia, abdominal fluid accumulation, and intra-abdominal infections, among others.

CONTACTS AND LOCATIONS:
Overall Officials: Shuo Jin, PhD, Principal Investigator — Beijing Tsinghua Chang Gung Hospital
Locations (1):
- Beijing Tsinghua Chang Gung Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No